CLINICAL TRIAL: NCT05174416
Title: A Phase III, Randomized, Double-blinded, Placebo-controlled Clinical Study With A Long-term Extension to Evaluate the Efficacy and Safety of Mavacamten in Chinese Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study to Evaluate the Efficacy and Safety of Mavacamten in Chinese Adults With Symptomatic Obstructive HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB2001-301
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
Keywords: Mavacamten
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mavacamten (Experimental): Mavacamten Capsules
  Interventions: Drug: Mavacamten
- placebo (Placebo Comparator): Matching Placebo Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavacamten — Mavacamten Capsules
  Other Names: MYK-461; BMS-986327
  Arms: Mavacamten
Drug: Placebo — Matching PBO capsules during placebo controlled period，and mavacamten capsules during long term extension period
  Arms: placebo

SUMMARY:
Mavacamtenis a novel, small molecule, selective allosteric inhibitor of cardiac-specific myosin, for the treatment of patients with symptomatic oHCM. This study will assess the efficacy and safety of mavacamten in Chinese adults with symptomatic oHCM.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled clinical study witha long-term extension to evaluate the efficacy and safety of mavacamten in Chinese adults with symptomatic oHCM. Approximately 81eligible participants will be enrolled and randomized in a 2:1 ratio (mavacamten:placebo). Participants will receive mavacamten or matching placebofor 30 weeks indouble-blinded manner. After 30-week double-blinded placebo-controlled treatment, eligible participants will receive mavacamten for additional 48 weeks (placebogroup: switch from placebo to mavacamten, mavacamten group: maintain on mavacamten).

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old at screening.
* Body weight is greater than 45 kg at screening.
* Has adequate acoustic windows to enable accurate TTEs
* Diagnosed with oHCM
* Has documented LVEF ≥ 55% at rest.
* Has a valid measurement of Valsalva LVOT peak gradient at screening
* Has NYHA Class II or III symptoms at screening
* Female participants must not be pregnant or lactating
* Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent according to national, local, and institutional guidelines before the first study specific procedure.

Exclusion Criteria:

* Participated in a clinical trial in which the participant received any investigational drug (or is currently using an investigational device) within 30 days prior to screening, or at least 5 times the respective elimination half-life (if known), whichever is longer.
* Causing cardiac hypertrophy in other reasons
* Previously participated in a clinical study with mavacamten.
* Hypersensitivity to any of the components of the mavacamten formulation.
* Current treatment (within 14 days prior to screening) or planned treatment during the double-blinded treatment with a combination of beta-blockers and verapamil or a combination of beta-blockers and diltiazem.
* Has been successfully treated with invasive septal reduction
* Has documented obstructive coronary artery disease
* Has known moderate or severe (as per investigator's judgment) aortic valve stenosis, constrictive pericarditis, or clinically significant congenital heart disease at screening.
* Has any acute or serious comorbid condition that, in the judgment of the investigator, could lead to premature termination of study participation or interfere with the measurement or interpretation of the efficacy and safety assessments in the study.
* History of malignant disease within 10 years of screening
* Has safety laboratory parameters outside normal limits at screening as assessed by the local laboratory
* Has a positive serologic test at screening for infection with human immunodeficiency virus, hepatitis C virus, or hepatitis B virus surface antigen.
* Known uncured COVID-19 (coronavirus disease 2019) infection or with severe complication before screening.
* Has a history or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Prior treatment with cardio toxic agents.
* Unable to comply with the study requirements, including the number of required visits to the clinical site.
* Is a first degree relative of personnel directly affiliated with the study at the clinical study site, any study vendor, or the study sponsor.
* Identified as alcohol addicts.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, M.D., Ph.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Z, Li L, Li X, Zhang Q, Peng D, Ma W, Yang P, Wang F, Cheng X, Fu Y, Sun J, Wang J, Zhang S. Effects of Mavacamten on Cardiac Magnetic Resonance Features in Chinese Patients With Obstructive Hypertrophic Cardiomyopathy. JACC Asia. 2025 Aug;5(8):1064-1074. doi: 10.1016/j.jacasi.2025.05.015. Epub 2025 Jul 8. PMID 40632050
- [Derived] Tian Z, Li X, Li L, Zhang Q, Wang J, Shi Y, Peng D, Yang P, Ma W, Wang F, Jin W, Cheng X, Chen YM, Zhong Y, Barrett YC, Zheng J, Zhang S. Effect of Mavacamten on Echocardiographic Features in Chinese Patients with Obstructive Hypertrophic Cardiomyopathy: Results from the EXPLORER-CN Study. Cardiol Ther. 2025 Jun;14(2):267-282. doi: 10.1007/s40119-025-00409-5. Epub 2025 Apr 29. PMID 40299193
- [Derived] Tian Z, Li L, Li X, Wang J, Zhang Q, Li Z, Peng D, Yang P, Ma W, Wang F, Jin W, Cheng X, Sun J, Fu Y, Lyu C, Zhang S. Effect of Mavacamten on Chinese Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy: The EXPLORER-CN Randomized Clinical Trial. JAMA Cardiol. 2023 Oct 1;8(10):957-965. doi: 10.1001/jamacardio.2023.3030. PMID 37639259
- [Derived] Tian Z, Wang F, Jin W, Zhang Q, Zhou J, Yang P, Wang G, Hsu P, Sun J, Zhang S, Han Y. Study design and rationale of EXPLORER-CN: a phase III, randomised, double-blind, placebo-controlled clinical study to evaluate the efficacy and safety of mavacamten in Chinese adults with symptomatic obstructive hypertrophic cardiomyopathy. BMJ Open. 2023 Jun 19;13(6):e071473. doi: 10.1136/bmjopen-2022-071473. PMID 37336533

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 81 eligible participants were randomly assigned to one of 2 treatment groups, mavacamten or placebo in a ratio of 2:1 (2 mavacamten and 1 placebo). Randomization was stratified according to current treatment at enrollment with a beta-blocker (yes or no)
Period: Overall Study
Arm/Group | Mavacamten | Placebo
Started | 54 | 27
Completed | 54 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavacamten | Placebo | Total
Number analyzed (Participants) | 54 | 27 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 23 | 70
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.08) | 51.0 (11.83) | 51.9 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 41 | 17 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 27 | 81
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 54 | 27 | 81
Valsalva LVOT peak gradient [Mean (Standard Deviation); unit: mmHg] | 106.78 (43.225) | 99.79 (41.100) | 104.45 (42.401)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 30 in Valsalva Left Ventricular Outflow Tract (LVOT) Peak Gradient
Description: To compare the effect of a 30-week course of mavacamten with placebo on Valsalva LVOT peak gradient as determined by Doppler echocardiography
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
mmHg | -51.05 (6.150) | 19.23 (8.535)

2. Secondary Outcome: Change From Baseline to Week 30 in Resting LVOT Peak Gradient
Description: To compare the effect of a 30-week course of mavacamten with placebo on LVOT obstruction.
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
mmHg | -49.04 (4.637) | 5.95 (6.311)

3. Secondary Outcome: Proportion of Participants Achieving a Valsalva LVOT Peak Gradient < 30 mmHg at Week 30
Description: To compare the effect of a 30-week course of mavacamten with placebo on LVOT obstruction.
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
Participants | 26 | 1

4. Secondary Outcome: Proportion of Participants Achieving a Valsalva LVOT Peak Gradient < 50 mmHg at Week 30.
Description: To compare the effect of a 30-week course of mavacamten with placebo on LVOT obstruction.
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
Participants | 32 | 2

5. Secondary Outcome: Proportion of Participants With at Least 1 Class Improvement in New York Heart Association (NYHA) Functional Classification From Baseline to Week 30
Description: To compare the effect of a 30-week course of mavacamten with placebo on clinical symptoms
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
Participants | 32 | 4

6. Secondary Outcome: Change From Baseline to Week 30 in Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS)
Description: To compare the effect of a 30-week course of Mavacamten with placebo on Participant-Reported health status individually The KCCQ (23-item version) is a patient-reported questionnaire that measures the impact of patients' CV disease or its treatment on 6 distinct domains using a 2-week recall: symptoms/signs, physical limitations, quality of life, social limitations, self-efficacy, and symptom stability (Green et al., 2000). In addition to the individual domains, 2 summary scores can be calculated from the KCCQ: the overall summary score (includes the total symptom, physical limitation, social limitations and quality of life scores) and the clinical summary score (combines the total symptom and physical limitation scales). Scores range from 0 to 100, with higher scores reflecting better health status. The KCCQ will be administered to participants as indicated.
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
score on a scale | 4.99 (2.063) | -5.25 (2.750)

7. Secondary Outcome: Change From Baseline to Week 30 in N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Description: To compare the effect of a 30-week course of mavacamten on cardiac biomarkers
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
ng/L | 0.182 (0.1743) | 0.932 (0.5133)

8. Secondary Outcome: Change From Baseline to Week 30 in Cardiac Troponin
Description: To compare the effect of a 30-week course of mavacamten on cardiac biomarkers
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
ng/L | 0.419 (0.1983) | 1.236 (0.6528)

9. Secondary Outcome: Change From Baseline to Week 30 in Left Ventricular (LV) Mass Index
Description: To compare the effect of a 30-week course of mavacamten with placebo on LV mass evaluated by cardiac magnetic resonance (CMR) imaging.
Time Frame: 30 weeks
Measure: Median (Standard Deviation); unit: g/m^2
Arm/Group | Mavacamten | Placebo
Number analyzed (Participants) | 54 | 27
g/m^2 | -26.365 (21.0565) | 4.434 (14.4226)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the first dose date of study medication up to 30 weeks.
Description: Consistent with clinicaltrials.gov definitions.
Arm/Group | Placebo | Mavacamten
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/27 | 4/54
Other Adverse Events (participants affected / at risk) | 24/27 | 45/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Mavacamten (N=54)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Mavacamten (N=54)
COVID-19 (Infections and infestations) | 11 | 20
Upper respiratory tract infection (Infections and infestations) | 4 | 8
Defect conduction intraventricular (Cardiac disorders) | 0 | 5
Palpitations (Cardiac disorders) | 2 | 3
Ventricular extrasystoles (Cardiac disorders) | 3 | 2
Cardiac discomfort (Cardiac disorders) | 0 | 3
Ventricular tachycardia (Cardiac disorders) | 2 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 4
Dizziness (Nervous system disorders) | 2 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 1
Hepatic enzyme increased (Investigations) | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 3
Hypertension (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT05174416/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT05174416/SAP_001.pdf